CLINICAL TRIAL: NCT06876480
Title: Evaluate of Different Visual Keyboard Organizations on People With Complex Sensorimotor Disabilities
Brief Title: Evaluation of Different Visual Keyboard Organizations on People With Complex Sensorimotor Disabilities
Acronym: SK4All
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP240703; 2024-A01067-40 (Registry Identifier: IDRCB)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Complex Sensorimotor Disabilities
Keywords: Complex sensorimotor disabilities; ScanningKeyboard

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm with virtual keyboard (Experimental): Arm with virtual keyboard: 16 days for each participant
  Interventions: Other: Keyboard

INTERVENTIONS:
Other: Keyboard — Day 0 : Collection of the general data required for the study, installation of the computer device including the LifeCompanion software with the different scanning keyboards configurations and organizations. Day 0 to Day 8 : write, in copy, a text using each of the virtual keyboard configurations. Day 8 : copying a text proposed by the investigator of identical difficulty for each condition, for a duration of 15 minutes, per experimental condition. This copying exercise, with the recording of measurements, will be done for each experimental condition. Day 8 to Day 16 : write a copy of a text of his/her choice for 10 minutes, using each of the virtual keyboard configurations. Day 16 : in a text-entry evaluation situation, copying a text proposed by the investigator, of identical difficulty for each condition.

SUMMARY:
comparison of different visual keyboard configurations

DETAILED DESCRIPTION:
Information and communication technologies (ICT) occupy an increasingly important place in our daily lives (CREDOC, 2021). Similarly, for the general population faced with these information and communication technologies, people with sensorimotor disabilities want and can claim socio-professional integration, access to knowledge through school integration facilitated by the Internet, access to leisure activities and social participation (Folan et al., 2015) (Picard, 2007) (Angelo et al., 2007) (Cornes & Bochel, 1987). Consequently, information and communication technologies are essential for people with sensorimotor disabilities and restoring this communication is fundamental.

Regarding access to digital tools, people with sensorimotor disabilities have difficulty accessing the pointing device (moving the mouse cursor, but also the various clicks) and input text (accessing the standard keyboard). Many assistive devices exist depending on the disabilities and abilities of the people, but also on their life habits, environmental constraints and expected uses of the computer tool (LoPresti and Brienza, 2004) (DeVries et al., 1998) (Yu-Luen Chen et al., 2003) (Y.-L. Chen et al., 2003) (Biard et al., 2011).

However, for people with complex sensorimotor disabilities, when few functional movements are possible, scanning access on a visual keyboard is preferred. At this stage, the movement of the mouse cursor, mouse clicks and text input are grouped under the same interface (visual keyboard) controlled by one or two switches. The visual keyboard presents the letters, the arrows for the direction of the mouse cursor and the different clicks (Figure 1).

In aims to increase people's text input speed, several studies have shown that the addition of linguistic prediction modules (of words or characters) would, in theory, make input text faster (Schadle & Poirier, 2004) (Trnka et al., 2007):

Word prediction (or completion) enables words or completions to be proposed in order to reduce the number of characters to be entered. By reducing the entry of certains characters, the text input speed should theoretically be increased. In fact, this is not necessarily the case (Raynal & Badr, 2022) (Pouplin et al., 2014).

Character prediction rearranges the layout of characters after each input, according to the probability of each one being selected. In this way, the most likely character becomes the one that can be accessed most quickly, with the least scanning. It has been shown that in the case of a pointing keyboard, this prediction does not satisfy users any more than word prediction (MacKenzie, 2008). Nevertheless, for scanning keyboards, which we are interested in here, even though there are few studies with real users, we can see that in some cases, character prediction seems interesting (Pouplin et al., 2014). Nevertheless, the main drawback of character prediction is that it results to a dynamic display of the keyboard. Indeed, the integration of character prediction seems to take place in much the same way from one study to the next, meaning a reorganization of the character set and therefore of the entire display. This prevents any memorization of the character layout for the user, and thus a certain amount of learning.

Therefore, we propose to integrate character prediction while keeping the display as static as possible.

ELIGIBILITY:
Inclusion Criteria:

* People with complex sensorimotor disabilities who are unable to communicate in standard written and digital form.
* Persons aged 18 or over
* Ability to read and write French
* Patient who own and use IT tool
* Patient who has used or used a virtual scanning keyboard to access IT Tools
* Health insurance beneficiary or rightful dependent
* Patient who has signed an informed and written consent. or
* Adult patient under guardianship who has signed an informed and written consent with the assistance of their guardian.
* Person agreeing to the terms of the protocol (home visits by the investigator).

Exclusion Criteria:

* Having visual impairments preventing the use of the IT Tools
* Patient under State Medical Aid (except in cases of exemption from affiliation).
* Persons deprived of liberty
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Text input speed evaluation | at 16 days
  To evaluate the influence of different visual keyboard organizations on text input speed in people with complex sensorimotor disabilities.
  Evaluation criteria: Text input speed (characters/minutes).

SECONDARY OUTCOMES:
Evaluate the influence of visual keyboard organizations on fatigue | at 16 days
  To evaluate the influence of different visual keyboard organizations on fatigue in people with complex sensorimotor disabilities.
  Evaluation criteria: Self-assessment of fatigue (Visual Analog Scale (VAS)).
Evaluation of usability efficiency | at 16 days
  To evaluate the influence of different visual keyboard organizations on the usability efficiency of the system by people with complex sensorimotor disabilities.
  Evaluation criteria: Input validity (percentage), System use strategy efficiency score (percentage).
Self-assessment of satisfaction | at 16 days
  To evaluaSelf-aste the influence of different visual keyboard organizations on text input system satisfaction in people with complex sensorimotor impairments.
  Self-assessment of satisfaction (Visual Analogue Scale (VAS)).
Oculometric data evaluation | at 16 days
  To evaluate the influence of different visual keyboard organizations on the distance covered by users' gaze.
  Evaluation criteria: Oculometric data (raw value).

CONTACTS AND LOCATIONS:
Overall Officials: SAMUEL POUPLIN, PhD, Principal Investigator — PFNT DEPARTMENT, Raymon Pincaré Hospital - APHP; Mathieu THEBAUD, Study Director — Laboratoire d'Assistances Technologiques, CMRRF Kerpape
Locations (1):
- CHU Raymond Poincaré - APHP, Garches, France

IPD SHARING:
Plan to Share IPD: No